CLINICAL TRIAL: NCT02080429
Title: Can Passive Descent Increase the Spontaneous Vaginal Delivery Rate in Obese Women?
Brief Title: Passive Descent in Obese Nulliparous Gravidae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Alisse Hauspurg, Resident Physician, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WIHRI-PD
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Management of the Second Stage of Labor in Obese Nulliparous Women by Either Passive Descent or Immediate Pushing.

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Pushing (Active Comparator): Patient's will begin to push when they are determined to be completely dilated.
  Interventions: Procedure: Pushing
- Passive Descent (Experimental): Patient's will wait 90 minutes prior to begin pushing
  Interventions: Procedure: Passive Descent

INTERVENTIONS:
Procedure: Passive Descent
  Arms: Passive Descent
Procedure: Pushing
  Arms: Immediate Pushing

SUMMARY:
Obesity rates in reproductive aged women in the United States are rising. It is now universally accepted that obesity is associated with many adverse pregnancy outcomes and post-operative complications following cesarean section. Recent studies have also shown an increased rate of cesarean section in obese women, adding to the already elevated rate of complications and adverse outcomes. Given the increased a priori risk for obese patients, it is vital that the investigators reexamine management practices routinely used for normal weight women in this specific high-risk population. Passive descent has been shown to increase the spontaneous vaginal delivery rate in non-obese women; however, high quality studies have never been performed in obese women. the investigators hypothesize that passive descent could improve the spontaneous vaginal delivery rate in nulliparous, obese women with regional anesthesia. This study will randomize women to passive descent for ninety minutes or active pushing upon entry into the second stage. Further, given that passive descent is widely accepted in the midwifery literature and clinical practice, the investigators anticipate that a high-quality study in the physician literature could increase the dialogue between practitioners and lead to development of best practices in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Obese - body mass index (BMI) calculated as weight (kg)/ [height (m2)] greater than or equal to 30 as determined at the time of admission to labor and delivery
* Regional anesthesia
* Nulliparous (defined as no deliveries after 20 weeks gestation)
* Gestational age of 37 0/7 weeks and greater
* Singleton Pregnancy

Exclusion Criteria:

* Body mass index (BMI) calculated as weight (kg)/ [height (m2)] less than 30 as determined at the time of admission to labor and delivery
* No regional anesthesia
* Multiparous
* Gestational age of less than 37 0/7 weeks
* Multiple gestations
* Maternal fever prior to second stage
* Severe fetal anomalies (incompatible with life)

Sex: Female
Age Groups: Child, Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Rate of spontaneous vaginal delivery | At delivery

SECONDARY OUTCOMES:
Rate of infections (defined as fever and / or antibiotic initiation) | participants will be followed for the duration of hospital stay, an expected average of 3 days
Rate of Third and Fourth Degree Lacerations | At delivery
Rate of Postpartum Hemorrhage | At delivery
Neonatal Outcomes | At delivery
  * admission to NICU
  * umbilical cord pH <7.1

CONTACTS AND LOCATIONS:
Overall Officials: Alisse Hauspurg, MD, Principal Investigator — Women & Infant's Hospital; Erika Werner, MD, Study Director — Women & Infant's Hospital
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States